CLINICAL TRIAL: NCT04370353
Title: Investigating the Impact of Cocoa Flavanol Supplementation on Pulmonary Oxygen Uptake Kinetics and Exercise Tolerance in Sedentary Middle-aged Adults
Brief Title: Impact of Cocoa Flavanols on Pulmonary Oxygen Uptake Kinetics and Exercise Tolerance in Sedentary Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 18/SPS/014
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Aging; Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo supplement, each capsule containing: 0mg total flavanols, matched for caffeine and theobromine content as experimental supplement (2.9 mg caffeine and 22.5 mg theobromine) and microcrystalline cellulose volume filler. Participants consume 4x capsules daily (2AM & 2PM after mixed meal for 7 days.
  Interventions: Dietary Supplement: Placebo supplement
- Cocoa Flavanols (Experimental): Experimental supplement, each capsule containing: 316 mg CocoActiv (Naturex, Netherlands: 100mg total cocoa flavanols, 2.9 mg caffeine and 22.5 mg theobromine) and microcrystalline cellulose volume filler. Participants consume 4x capsules daily (2AM & 2PM) for 7 days.
  Interventions: Dietary Supplement: Cocoa flavanols

INTERVENTIONS:
Dietary Supplement: Cocoa flavanols — Flavonoid-rich cocoa powder, containing 100mg total flavanols per 316mg.
  Arms: Cocoa Flavanols
Dietary Supplement: Placebo supplement — Microcrystalline filler, containing 0mg total flavanols.
  Arms: Placebo

SUMMARY:
In recent years, there has been significant interest in dietary flavonoids (biologically active plant-derived compounds) as potential therapeutics. This is due to the capacity of flavonoids to enhance processes related to energy metabolism and cardiovascular health. We are interested in implementing a short-term supplementation regime (daily cocoa-flavanoid ingestion), in order to explore the possible beneficial effects of flavonoid-based interventions on responses to exercise. Hence, the objective of our study is to examine the impact of short term cocoa-flavanoid supplementation on processes related to energy use (oxygen utilisation). Our aim is to develop a novel intervention which improves cardiovascular health and enhances exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-55 years
* Healthy (no known cardiovascular or metabolic disorders e.g. diabetes)
* Do not engage in regular structured physical training (i.e. less than two sessions for 60 minutes per week, for at least 1 year

Exclusion Criteria:

* Smokers
* Medical history of cardiovascular and/or metabolic disease, including diabetes and abnormal blood pressure
* Family history of cardiovascular disease
* Currently taking any medication
* Asthmatic
* Currently suffering from musculoskeletal injury
* Younger than 35 or older than 55 years old
* Known food allergies or special dietary requirements
* Currently taking any dietary supplements
* Currently engaging in >2 hours structured training per week

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake kinetics | Over 3 week period (After 7 days of each intervention). Oxygen uptake measured for 9 minutes continuously during exercise bouts (3 min warm up period and 6 minutes of exercise transition)
  Oxygen uptake kinetics (including time constant, time delay and amplitude of the fundamental oxygen uptake response) will be determined by modelling oxygen uptake during exercise using a mono exponential function. The oxygen uptake data is measured on a breath-by-breath basis during exercise (on a cycle ergometer) using a gas analysis system and face mask. Oxygen kinetics will be measured during three moderate-intensity step exercise tests (at 80% of the gas exchange threshold) and during one severe-intensity (60%∆) step exercise test that is completed to failure.
Exercise tolerance | Over 3 week period (After 7 days of each intervention).
  Participants capacity to exercise to the limit of tolerance, measured to the nearest second. Participants are instructed to exercise at a severe-intensity exercise load (representative of 60% ∆), on a cycle ergometer until volitional exhaustion.

SECONDARY OUTCOMES:
Heart rate | Over 3 week period (After 7 days of each intervention). Measured during the length of each exercise transition (9 minutes for each moderate intensity bout).
  Heart rate will be measured during moderate and severe-intensity exercise bouts, by short-range telemetry.
Blood pressure | Over 3 week period (After 7 days of each intervention). Measured over 5 minutes before any exercise testing.
  Systolic and diastolic blood pressure will be assessed following 10 min of seated rest using an automated sphygmomanometer
Blood lactate | Over 3 week period (After 7 days of each intervention). Measured immediately before and after exercise
  A finger prick blood sample will be taken to measure blood lactate pre- and post-exercise of each transition using a hand-held automated blood lactate analyser
Physical activity and sedentary behaviour | Over 3 week period (In the 6 days preceding experimental testing)
  Physical activity levels will be assessed in the 6 days prior to visiting the laboratory by an accelerometer, worn on the hip during waking hours.
Perceived workload | Over 3 week period (After 7 days of each intervention). Measured immediately before and after exercise
  Perceived mental workload will be measured pre and post exercise using NASA Task Load Index and BORG rating of perceived exertion scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Sport & Exercise Sciences, Liverpool, United Kingdom

REFERENCES:
- [Derived] Sadler DG, Draijer R, Stewart CE, Jones H, Marwood S, Thijssen DHJ. Cocoa-flavanols enhance moderate-intensity pulmonary V O 2 kinetics but not exercise tolerance in sedentary middle-aged adults. Eur J Appl Physiol. 2021 Aug;121(8):2285-2294. doi: 10.1007/s00421-021-04682-9. Epub 2021 May 10. PMID 33970327